CLINICAL TRIAL: NCT00371540
Title: Extending HIV Care Beyond the Rural Health Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Moi Univeristy (Other)
Responsible Party: Principal Investigator, Kara Wools-Kaloustian, Associate Professor, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DDCF 2005043
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-11

CONDITIONS: HIV; HIV Infections
Keywords: Africa; Antiretrovirals
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (No Intervention): Routine care in the clinic
- II (Experimental): Follow-up in clinic every 3 months, home visits monthly
  Interventions: Other: Home visit by community care coordinators

INTERVENTIONS:
Other: Home visit by community care coordinators — Decrease in patient visits to the clinic from the standard of once per month to every 3 months with home visits monthly.
  Arms: II

SUMMARY:
The objective of this application is to develop and assess a system which uses non-clinician extenders to provide selected aspects of HIV care in rural western Kenya. The plan is to train persons living with HIV/AIDS (PLWAs) to undertake this role as Community Care Coordinators. Our central hypothesis, is that PLWAs can be effective members of the health care team and that their involvement in community-based HIV care will facilitate patient access to services and improve outcomes. As such our two specific aims are: 1) To develop a sustainable system to extend HIV care into the community and to train the individuals necessary to support such a system (Community Care Coordinators). 2) To determine the impact of Community Care Coordinators on patient adherence (to drugs and to clinic visits), clinical outcomes (i.e. viral load responses [an individuals level of circulating HIV virus], inter-current opportunistic infections, hospitalization, drop out from the program, change to second line therapy and mortality) and patient perception of stigma. This study will provide invaluable data on the use of non-clinician care extenders for providing HIV care in resource poor settings. As such, knowledge gained from this study will assist in developing a model for non-clinician centered HIV care systems elsewhere in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infected
2. >18 years old
3. household members are aware of the patient's HIV infection
4. clinically stable on ARVs and no significant adherence issues for 3 months, 5) live in Kosirai Division

6) willing to consent to participate.

Exclusion Criteria:

1. active opportunistic infection
2. pregnant
3. hospitalized in the previous 3 months
4. unable to understand the informed consent process due to mental or physical incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara K Wools-Kaloustian, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Mosoriot Rural Health Center, Mosoriot, Kenya

REFERENCES:
- [Derived] Selke HM, Kimaiyo S, Sidle JE, Vedanthan R, Tierney WM, Shen C, Denski CD, Katschke AR, Wools-Kaloustian K. Task-shifting of antiretroviral delivery from health care workers to persons living with HIV/AIDS: clinical outcomes of a community-based program in Kenya. J Acquir Immune Defic Syndr. 2010 Dec;55(4):483-90. doi: 10.1097/QAI.0b013e3181eb5edb. PMID 20683336
- [Derived] Wools-Kaloustian KK, Sidle JE, Selke HM, Vedanthan R, Kemboi EK, Boit LJ, Jebet VT, Carroll AE, Tierney WM, Kimaiyo S. A model for extending antiretroviral care beyond the rural health centre. J Int AIDS Soc. 2009 Sep 29;12:22. doi: 10.1186/1758-2652-12-22. PMID 19788755

RESULTS

PARTICIPANT FLOW:
Groups:
- I Routine Care: Routine care in the clinic
- II Home Visits: Follow-up in clinic every 3 months, home visits monthly
  Home visit by community care coordinators: Decrease in patient visits to the clinic from the standard of once per month to every 3 months with home visits monthly.
Period: Overall Study
Arm/Group | I Routine Care | II Home Visits
Started | 112 | 96
Completed | 102 | 87
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Population: HIV infected patients who were clinically stable on ART for at least 3 months
Groups:
- Total: Total of all reporting groups
Arm/Group | I Routine Care | II Home Visits | Total
Number analyzed (Participants) | 112 | 96 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 96 | 208
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 81 | 71 | 152
  Male | 31 | 25 | 56
Region of Enrollment [Number; unit: participants]
  Kenya | 112 | 96 | 208

OUTCOME MEASURES:

1. Secondary Outcome: Viral Load
Description: Detectable VL at 12 months
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | I Rountine Care | II Home Visits
Number analyzed (Participants) | 96 | 86
participants | 13 | 9
Statistical Analysis 1: Comparison: I Rountine Care vs II Home Visits; Note: The differences between the number of individuals evaluable for this secondary outcome and the number of individuals evaluable for the primary outcome is related to specimen loss by the laboratory. As such of the Routine care group only 96 of 102 patients completing the study were evaluable for the viral load outcome and only 86 of 87 patients in the Home visit group; Test type: Superiority or Other; p = 0.65, Fisher Exact

2. Primary Outcome: Lost to Follow-up
Description: Number of Subjects Lost to follow-up
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | I Rountine Care | II Home Visits
Number analyzed (Participants) | 112 | 96
participants | 5 | 5
Statistical Analysis 1: Comparison: I Rountine Care vs II Home Visits; Test type: Superiority or Other; p = 1.0, Fisher Exact

3. Secondary Outcome: Death
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | I Rountine Care | II Home Visits
Number analyzed (Participants) | 112 | 96
participants | 0 | 1
Statistical Analysis 1: Comparison: I Rountine Care vs II Home Visits; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | I Rountine Care | II Home Visits
Serious Adverse Events (participants affected / at risk) | 0/112 | 1/96
Other Adverse Events (participants affected / at risk) | 0/112 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I Rountine Care (N=112) | II Home Visits (N=96)
Death (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Patient self prescribed and administered an herbal Abortifacient precipitating hemorrhage and death. This death was not related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No